CLINICAL TRIAL: NCT05396469
Title: Using Thoracic Ultrasound in a Rheumatological Setting to Detect Interstitial Lung Disease in Patients With Rheumatoid Arthritis: Protocol for a Cross-Sectional Diagnostic Test Accuracy Study. AURORA.
Brief Title: Using Thoracic Ultrasound to Detect Interstitial Lung Disease in Patients With Rheumatoid Arthritis
Acronym: AURORA
Status: Completed | Type: Observational
Sponsor: Torkell Ellingsen (Other)
Responsible Party: Sponsor-Investigator, Torkell Ellingsen, MD, PhD, Clin. Professor, Consultant, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: S-20210154
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis and Associated Conditions; Lung Diseases, Interstitial
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: National guideline treatment — All discovered diseases will recieve national guideline treatment and follow up

SUMMARY:
Background: Pulmonary diseases are significant contributors to morbidity and mortality in patients with rheumatoid arthritis (RA). One of the most common pulmonary manifestation in RA is interstitial lung disease (RA-ILD). Consequently, RA-ILD may be prevalent in approximately 30% and clinically evident in about 10% of RA patients. Since the median survival for patients with manifest RA-ILD is only 6.6 years, feasible methods of detecting early RA-ILD are warranted.

Objectives: To determine the diagnostic accuracy of thoracic ultrasound (TUS), using a 14-zone protocol, for ILD in RA patients with respiratory symptoms by using chest high-resolution computed tomography (HRCT) as the reference standard. The secondary aim is to evaluate the diagnostic accuracy for the blood biomarkers surfactant protein-D (SP-D) and microfibrillar-associated protein 4 (MFAP4) in the detection of ILD in this group of patients.

Data collection: Participants will be included after signing the informed consent; data will be collected and stored in a REDCap database.

Eligibility criteria for participants and settings where data will be collected: Patients eligible for inclusion are consenting adults (≥18 years) diagnosed with RA (according to the 2010 ACR-criteria for RA) and respiratory symptoms indicating RA-ILD, based on the presence of at least one of the following symptoms: unexplained dyspnoea, unexplained cough and/or a residual pneumonia or a chest X-ray indicating interstitial abnormalities in the lung.

Whether participants form a consecutive, random or convenience series: Participants form a consecutive series of up to 80 individuals in total.

Description of the index test and reference standard: Patients suspected of having RA-ILD will undergo a 14 zone TUS as index test performed by a junior resident in rheumatology, who is certified by the European Respiratory Society in performing TUS assessment. The anonymised images will be stored, and scored by the junior resident and two senior rheumatologists, who have also received training in TUS, as well as a TUS and ILD experienced pulmonologist. Chest HRCT will be the gold standard, i.e. the ILD reference standard.

Estimates of diagnostic accuracy and their precision: The two basic measures for quantifying the diagnostic accuracy of the TUS (index) test are the sensitivity and specificity in comparison to the chest HRCT. Statistical tests will be conducted using the McNemar test for correlated proportions.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion are consenting adults (≥18 years) diagnosed with RA, with presence of at least one of the following symptoms: unexplained dyspnoea, unexplained cough, residual pneumonia or a chest X-ray indicating interstitial lung disease. All patients must fulfil the 2010 criteria for RA. A diagnosis of COPD does not exclude the patient from the study.

Exclusion Criteria:

* Patients with other systemic autoimmune diseases than RA (except secondary Sjøgrens syndrome) will be excluded. Other exclusion criteria are; previous or active lung cancer, lung transplant recipients and patients with known ILD or congenital lung disease, as well as patients who have had an HRCT performed within 12 months prior to the inclusion date. Patients who are unwilling or unable to provide written informed consent will also be excluded (i.e. not eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited from the Department of Rheumatology in the Hospital of South West Jutland, Odense University Hospital - Svendborg Hospital, Lillebaelt Hospital and Odense University Hospital (OUH). Patients coming inn for a planned control of their RA disease and management, will be asked if they have respiratory symptoms. If respiratory symptoms are present, the patient will receive oral information about this project and those who are interested in participating, will receive written information as well as a signed consent form (not yet to be signed). Subsequently, the patients will be referred to the highly specialized unit in the Department of Rheumatology at OUH as well as a full clinical evaluation in the PUlmo-REuma (PURE) Clinic located at OUH.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
RA-ILD | 31.01.2024
  Estimates of diagnostic accuracy and precision: The diagnostic accuracy of the TUS (index) test for interstitial lung disease in rheumatoid arthritis in comparison to the chest HRCT.

CONTACTS AND LOCATIONS:
Overall Officials: Torkell Ellingsen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Rheumatology Research Unit, Dept. of Rheumatology, OUH, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from the AURORA study will be stored in the Danish Data Archive (DDA) when data have been analysed and published. Through an agreement with the Danish Data Protection agency, the DDA preserves data materials containing personal identifiers. Data and the personal identifiers will be stored separately and special permits are required for access to the data. Data will be available on request for academic researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 31.01.2024 - 31.01.2034
Access Criteria: Data will be available on request for academic researchers.

REFERENCES:
- [Derived] Sofiudottir BK, Harders S, Laursen CB, Lage-Hansen PR, Nielsen SM, Just SA, Christensen R, Davidsen JR, Ellingsen T. Detection of Interstitial Lung Disease in Rheumatoid Arthritis by Thoracic Ultrasound: A Diagnostic Test Accuracy Study. Arthritis Care Res (Hoboken). 2024 Sep;76(9):1294-1302. doi: 10.1002/acr.25351. Epub 2024 Jun 23. PMID 38622106
- [Derived] Sofiudottir BK, Harders SMW, Lage-Hansen PR, Christensen R, Munk HL, Sorensen GL, Davidsen JR, Ellingsen T. Using thoracic ultrasound to detect interstitial lung disease in patients with rheumatoid arthritis: a protocol for the diagnostic test accuracy AURORA study. BMJ Open. 2022 Dec 23;12(12):e067434. doi: 10.1136/bmjopen-2022-067434. PMID 36564119